CLINICAL TRIAL: NCT02891863
Title: Low Energy Therapy Application to Convert Ventricular Tachycardias (LEVER)
Brief Title: Low Energy Therapy to Convert Ventricular Tachycardias
Acronym: LEVER
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Futility
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91003730
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2016-08

CONDITIONS: Ventricular Tachycardia
Keywords: Implantable Cardioverter-Defibrillator
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute Testing (Experimental): Single-arm study - all subjects who meet the I&E criteria, sign the consent form and have inducible VT within the protocol-specified criteria may be tested for VT conversion with the LEVER Acute Study System.
  Interventions: Device: LEVER Acute Study System

INTERVENTIONS:
Device: LEVER Acute Study System — The LEVER Acute Study System is an acute pacing and shock delivery system intended for investigational use only. The LEVER Acute Study System is intended for acute conversion testing of monomorphic ventricular tachycardia by one of three different VT conversion methods.

SUMMARY:
The LEVER study is a prospective, unblinded, non-randomized, first in human feasibility study that will assess and characterize early safety and effectiveness of low energy therapies in converting monomorphic ventricular tachycardias (MVTs).

DETAILED DESCRIPTION:
The LEVER study is a prospective, unblinded, non-randomized, first in human feasibility study that will assess and characterize early safety and effectiveness of low energy therapies in converting monomorphic ventricular tachycardias (MVTs). Subjects must be already indicated for standard of care VT procedure during which VT is likely to be induced (such as VT testing, VT ablation, VT mapping, or VT risk stratification testing.)

The study patches will be applied to the subject's torso, and the patches will be connected to the LEVER Acute Study System. Pacing capture threshold capture may be assessed. If monomorphic VT is induced and reaches at least 170bpm (350ms/cycle), one or more of the low energy therapies will be applied under oversight of the investigator, in an attempt to treat and convert the VT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of ventricular tachycardia indicated for ventricular testing procedures that may include VT induction, such as VT testing, VT ablation, VT mapping, or VT risk stratification testing.
* Subjects age 18 or above, or of legal age to give written informed consent specific to local laws and requirements
* Subjects who, in the opinion of the investigator, are suitable to be enrolled in a clinical study

Exclusion Criteria:

* Subjects with any comorbidities that, in the opinion of the investigator, would exclude them from standard of care VT testing
* Subjects with VT that is known to be focal in nature
* Subjects whom the investigator believes are not hemodynamically stable enough to tolerate testing
* Subjects of childbearing age who may be pregnant.
* Subjects who are unwilling or unable to provide written informed consent.
* Subjects with any implanted device that emits electrical energy where either therapy cannot be temporarily disabled, or the subject cannot tolerate temporary disabling of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Roberts-Thompson, MD, Principal Investigator — Royal Adelaide Hospital; Andreas Bollmann, MD, Principal Investigator — Hertz Centrum, Leipzig
Locations (1):
- Royal Adelaide Hospital, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No
Acute feasibility study of possible new product feature, confidential information

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acute Testing
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acute Testing
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: System and Procedure Related Adverse Events
Description: All system and procedure-related adverse events through 7 days (-1/+3 days) post-procedure will be collected and tracked.
Time Frame: 7 days post-procedure
Measure: Number; unit: participants
Arm/Group | Acute Testing
Number analyzed (Participants) | 9
participants | 5

2. Primary Outcome: Conversion Efficacy of Low Energy VT Therapies
Description: Effectiveness of LEVER Acute Study System low energy therapies to convert MVTs will be collected and tracked as an aggregate success rate (%) on a per-attempt basis for each therapy tested.
Time Frame: Acute - eg within 5 seconds of test therapy delivery
Population: 6 of 9 subjects had at least one inducible VT, a total of 14 attempts to convert VT with multiple pulses were delivered and none converted the VT in any subject.
Measure: Number; unit: percentage of VF conversion success
Units Other Than Participants: Attempts at VF Conversion
Arm/Group | Acute Testing
Number analyzed (Participants) | 6
Number analyzed (Attempts at VF Conversion) | 14
percentage of VF conversion success | 0

ADVERSE EVENTS:
Time Frame: from the time of the acute testing until 7 days post-procedure
Arm/Group | Acute Testing
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Testing (N=9)
post-procedure VT recurred (Cardiac disorders) | 1 (1) — patient had a recurrence of VT post-procedure (likely due to unsuccessful VT ablation that was not a specific aspect of the study)
VT accelerated to VF (Cardiac disorders) | 1 (1) — during the procedure an induced VT accelerated to VF, but was successfully converted. This is not unexpected for a such a procedure involving VT induction.
LV impairment (Cardiac disorders) | 1 (1) — 7 days post-procedure the pt had chest pain, and was found to have LV impairment. The condition resolved and the subject was released 2 days later.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acute Testing (N=9)
muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1) — pt temporarily reported muscle soreness after the procedure
VT acceleration to VF (Cardiac disorders) | 1 (1) — during the procedure a VT spontaneously occurred that accelerated to VF and was converted by an external shock

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This an early-stage feasibility study with significant intellectual property value to the sponsor. The sponsor controls access to the data and no publications can be submitted without the sponsors approval. Since the study was stopped early due to futility it may not be publishable, but preliminary data was submitted via abstract for presentation at Heart Rhythm 2017.